CLINICAL TRIAL: NCT02147951
Title: A Phase 3b, Multicenter, Open-label, Single-arm, Expanded Access Protocol of Talimogene Laherparepvec for the Treatment of Subjects With Unresected, Stage lllB to IVM1c Melanoma
Brief Title: Expanded Access Protocol of Talimogene Laherparepvec for Subjects With Unresected, Stage lllB to IVM1c Melanoma
Status: No longer available | Type: Expanded Access
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20120166
Record Dates: First submitted 2014-05-01; First posted 2014-05-28 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Unresected Stage IIIb to IVM1c Melanoma
Keywords: Melanoma
MeSH Terms: conditions — Melanoma | interventions — talimogene laherparepvec

INTERVENTIONS:
Drug: Talimogene Laherparepvec — Up to 4ml of talimogene laherparepvec per cycle visit

SUMMARY:
Expanded access of Talimogene Laherparepvec for subjects with unresected, stage IIIb to IVM1c Melanoma.

DETAILED DESCRIPTION:
Expanded access of Talimogene Laherparepvec for subjects with unresected, stage IIIb to IVM1c Melanoma that may not meet the eligibility criteria to enroll in another ongoing Talimogene Laherparepvec study or do not have access to enroll in an ongoing Talimogene Laherparepvec study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of melanoma
* Subject has unresected stage lllB to IVM1c melanoma regardless of prior therapy
* Subject who is not eligible for or cannot access ongoing talimogene laherparepvec clinical trials
* Candidate for intralesional therapy (ie, disease is appropriate for direct injection or through the use of ultrasound guidance) defined as one of the following:
* for a subject not previously treated with talimogene laherparepvec:
* at least 1 injectable cutaneous, subcutaneous, or nodal melanoma lesion ≥ 10 mm in longest diameter, or
* multiple injectable melanoma lesions that in aggregate have a longest diameter of ≥ 10 mm
* for a subject previously treated with talimogene laherparepvec:
* at least 1 injectable cutaneous, subcutaneous, or nodal melanoma lesion must be present (no minimal size criteria)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Adequate organ function determined within 35 days prior to enrollment
* Serum LDH levels less than or equal to 1.5 ULN within 35 days prior to enrollment
* For a subject who previously received talimogene laherparepvec in another clinical trial, subject must have ended treatment for reason(s) other than disease progression or intolerability to talimogene laherparepvec

Exclusion Criteria:

* Clinically active cerebral metastases. Subjects with up to 3 (neurological performance status of 0) cerebral metastases may be enrolled, provided that all lesions have been adequately treated with stereotactic radiation therapy, craniotomy, gammaknife therapy, with no evidence of progression, and have not required steroids, for at least two (2) months prior to enrollment.
* Greater than 3 visceral metastases (this does not include lung metastases or nodal metastases associated with visceral organs). For subjects with less than or equal to 3 visceral metastases, no lesion > 3 cm, and liver lesions must meet RECIST criteria for stable disease for at least 1 month prior to enrollment.
* Bone metastases
* Primary ocular or mucosal melanoma
* History or evidence of symptomatic autoimmune pneumonitis, glomerulonephritis, vasculitis, or other symptomatic autoimmune disease
* Evidence of clinically significant immunosuppression
* Active herpetic skin lesions or prior complications of HSV-1 infection (eg, herpetic keratitis or encephalitis)
* Requires intermittent or chronic systemic (intravenous or oral) treatment with an antiherpetic drug (eg, acyclovir), other than intermittent topical use
* Currently receiving treatment with another investigational device or drug study besides talimogene laherparepvec, or less than 28 days since ending treatment with another investigational device or drug study(s)
* Other investigational procedures while participating in this protocol are excluded
* Known to have acute or chronic active hepatitis B or hepatitis C infection
* Known to have human immunodeficiency virus infection
* History of other malignancy within the past 3 years with the following exceptions:
* malignancy treated with curative intent and with no known active disease present for ≥ 3 years before enrollment and felt to be at low risk for recurrence by the treating physician
* adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
* adequately treated cervical carcinoma in situ without evidence of disease
* adequately treated breast ductal carcinoma in situ without evidence of disease
* prostatic intraepithelial neoplasia without evidence of prostate cancer
* adequately treated urothelial papillary noninvasive carcinoma or carcinoma in situ
* Subject has known sensitivity to any of the products or components to be administered during dosing
* History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator or Amgen medical monitor, if consulted, would pose a risk to subject safety or interfere with the protocol evaluation, procedures or completion
* Female subject is pregnant or breast-feeding, or planning to become pregnant during protocol treatment and through 3 months after the last dose of talimogene laherparepvec
* Female subject of childbearing potential who is unwilling to use acceptable method(s) of effective contraception during protocol treatment and through 3 months after the last dose of talimogene laherparepvec

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (21):
- United States (21):
  - Research Site, Mobile, Alabama
  - Research Site, Little Rock, Arkansas
  - Research Site, Duarte, California
  - Research Site, La Jolla, California
  - Research Site, Daytona Beach, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami Beach, Florida
  - Research Site, Indianapolis, Indiana
  - Research Site, Louisville, Kentucky
  - Research Site, Minneapolis, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, Morristown, New Jersey
  - Research Site, New York, New York
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Canton, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Greenville, South Carolina
  - Research Site, Dallas, Texas
  - Research Site, Franklin, Wisconsin
  - Research Site, Wauwatosa, Wisconsin

REFERENCES:
- [Derived] Chesney J, Imbert-Fernandez Y, Telang S, Baum M, Ranjan S, Fraig M, Batty N. Potential clinical and immunotherapeutic utility of talimogene laherparepvec for patients with melanoma after disease progression on immune checkpoint inhibitors and BRAF inhibitors. Melanoma Res. 2018 Jun;28(3):250-255. doi: 10.1097/CMR.0000000000000444. PMID 29561296
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com